CLINICAL TRIAL: NCT02184325
Title: Safety and Tolerability of Kiddi® Pharmaton Fizz Effervescent Tablets, Comparing the Marketed Formula With an Improved One With a Reduced Mineral Amount, and a Comparator Product: a Double-blind, Controlled, Randomised, Three Arm Cross-over Study in Children
Brief Title: Safety and Tolerability of Kiddi® Pharmaton Fizz Effervescent Tablets in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1129.2
Record Dates: First submitted 2014-07-08; First posted 2014-07-09 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (3):
- Kiddi® Pharmaton Fizz, effervescent tablets (Experimental): with reduced amount of minerals
  Interventions: Drug: Kiddi® Pharmaton Fizz, effervescent tablets
- Kiddi® Pharmaton Fizz, effervescent tablets: marketed formula (Active Comparator)
  Interventions: Drug: Kiddi® Pharmaton Fizz, effervescent tablets: marketed formula
- Comparator product (Active Comparator): in the form of a product that is a market leader
  Interventions: Drug: Comparator product

INTERVENTIONS:
Drug: Kiddi® Pharmaton Fizz, effervescent tablets
  Arms: Kiddi® Pharmaton Fizz, effervescent tablets
Drug: Kiddi® Pharmaton Fizz, effervescent tablets: marketed formula
  Arms: Kiddi® Pharmaton Fizz, effervescent tablets: marketed formula
Drug: Comparator product — active substances: Vitamin A, Vitamin B1, Vitamin B2, Vitamin B5, Vitamin B6, Vitamin B12, Vitamin C, Vitamin D, Vitamin E, Manganese, Copper, Calcium, Magnesium, Phosphorous, Iron, Zinc, Sodium, Molybden
  Arms: Comparator product

SUMMARY:
Study to evaluate the tolerability and safety of Kiddi® Pharmaton Fizz effervescent tablets, in children of 6 to 14 years, comparing a given formula with an improved one with reduced mineral content (qualitatively equivalent to the first one) and a comparator product.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes aged between 6 and 14 years, inclusive
* Children, healthy or during convalescence, for which prevention or treatment of marginal vitamin deficits is indicated
* Willingness of the children and parents to give their written informed consent, according to Good Clinical Practice and local regulations
* Pregnant children will not be excluded

Exclusion Criteria:

* Has taken medications containing vitamins A or D, retinoids, or iron during the 4 weeks preceding the study enrolment
* Pre-treatment (less than 2 weeks prior the inclusion in this trial) and/or concomitant treatment with any drug that may influence the trial symptomatology, and may interfere with the evaluation of the safety of the test drug
* Participation in other clinical trials within the last 4 weeks and concurrent participation in another clinical trial
* Relevant allergy or kown hypersensitivity to one of the ingredients of the investigational drug
* Has any serious disorder that may interfere with the participation to the trial
* Malabsorption syndrome, liver and/or renal diseases or juvenile diabetes
* Increased calcium blood concentration, or an increased calcium-excretion
* Evident states of protein deficiency
* Presence of lysinemia (defect of the enzyme lysine ketoglutarate reductase)

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 1999-11; Primary Completion 2000-02 (Actual)

PRIMARY OUTCOMES:
Incidence of total drug-related adverse events | up to 19 days

SECONDARY OUTCOMES:
Incidence of all individual drug-related adverse events | up to 19 days
Assessment of overall tolerability and acceptance on a 4-point verbal rating scale | up to day 19